CLINICAL TRIAL: NCT03307200
Title: A Prospective Observational Study on the Unmet Supportive Care Needs of Bladder Cancer Patients Undergoing Radical Cystectomy
Brief Title: Unmet Supportive Care Needs in Bladder Cancer Patients Undergoing Radical Cystectomy
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Other Study IDs: EC/2017/0350
Record Dates: First submitted 2017-09-22; First posted 2017-10-11 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Bladder Cancer; Urologic Cancer; Surgery
Keywords: Supportive care; Prospective observational study
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Nowadays, high-quality cancer care is more than just diagnosis and treatment of cancer. Healthcare must respond to the specific needs of the patients to provide patient-centered care. To date, research on the unmet supportive care needs in bladder cancer patients undergoing radical cystectomy is scarce. Because the needs of the patients may differ according to the phase in the illness trajectory, it is important that prospective research is carried out. Research in other cancer populations shows that unmet supportive care needs are negatively associated with health-related quality of life, psychological distress, physical activity and the health literacy of the patient. By incorporating the above factors into this study, we can not only map the unmet supportive care needs of the patient, but also explore possible associations between the variables. Since this is the first prospective study on supportive care needs in bladder cancer, this is a hypothesis-generating study.

ELIGIBILITY:
Inclusion Criteria:

* age is 18 years or older
* Patients diagnosed with bladder cancer who will undergo radical cystectomy
* Patient has to be able to sign informed consent

Exclusion Criteria:

* Metastatic cancer
* Presence of a second primary tumor with the exception of fully deleted prostate cancer, non-melanoma skin tumor or tumor diagnosed ≥ 5 years ago and under control

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with bladder cancer who will undergo radical cystectomy
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Change in Unmet supportive care needs | From baseline up to 1 year
  Assessed with the 34-item supportive care needs survey (SCNS-34)

SECONDARY OUTCOMES:
Change in Cancer-specific Health-related quality of life | From baseline up to 1 year
  Assessed with the EORTC-qlq-c30
Change in Bladder cancer-specific Health-related quality of life | From baseline up to 1 year
  Assessed with the EORTC-qlq-blm30
Change in Psychological distress | From baseline up to 1 year
  Assessed with the distress thermometer
Change in problems associated with psychological distress | From baseline up to 1 year
  Assessed with the problem list
Health literacy | Baseline
  Assessed with the BRIEF Health Literacy Screening Tool
Change in Physical activity pattern | From baseline up to 1 year
  Assessed with the Godin Leisure-Time Exercise Questionnaire
Change in Physical Activity Stage of change | From baseline up to 1 year
  Assessed with a questionnaire based on an algorithm made by Marcus et al.
Change in The use of health care services | From baseline up to 1 year
  Separate questions where the patient is asked about his/her use of supportive health care services.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Fonteyne, MD, PhD, Principal Investigator — Gent University
Locations (2):
- Belgium (2):
  - Ghent University, Ghent
  - University Hospitals Leuven, Leuven

REFERENCES:
- [Derived] Rammant E, Van Hecke A, Decaestecker K, Albersen M, Joniau S, Everaerts W, Jansen F, Mohamed NE, Colman R, Van Hemelrijck M, Fonteyne V. Supportive care needs and utilization of bladder cancer patients undergoing radical cystectomy: A longitudinal study. Psychooncology. 2022 Feb;31(2):219-226. doi: 10.1002/pon.5795. Epub 2021 Aug 27. PMID 34449941